CLINICAL TRIAL: NCT05857085
Title: Impact of Additional Treatment With Empagliflozin or Semaglutide on Endothelial Function and Other Clinical Parameters and Biomarkers in T1DM Patients
Brief Title: Novel Therapeutics and Endothelial Dysfunction in T1DM Patients
Acronym: ENDIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: General and Teaching Hospital Celje (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-63-2020
Record Dates: First submitted 2020-09-29; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Endothelial Dysfunction; Diabetes Mellitus, Type 1; Biomarkers; Endothelial Progenitor Cells; SGLT 2 Inhibitors; Incretins; Glucose Excursions; FMD; FPF; Arterial Stiffness
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — semaglutide; empagliflozin

STUDY DESIGN:
Intervention Model Description: 2 therapeutic arms - adding empagliflozin or semaglutide to basic insulin treatment and control arm in type 1 diabetic patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GLP 1 agonist (Active Comparator): semaglutide in titrating doses 0,25 to 1,0 mg - duration of treatment12 weeks adding to insulin sheme (MDI or CII)
  Interventions: Drug: Semaglutide Pen Injector [Ozempic]
- SGLT 2 inhibitor (Active Comparator): empagliflozin 25 mg - duration of treatment 12 weeks adding to insulin sheme (MDI or CII or hybride system)
  Interventions: Drug: Empagliflozin 10 MG
- comparator (No Intervention): continuing treatment only with insulin sheme (MDI or CII or hybride system)

INTERVENTIONS:
Drug: Semaglutide Pen Injector [Ozempic] — GLP 1 agonist
  Arms: GLP 1 agonist
Drug: Empagliflozin 10 MG — SGLT 2 inhibitor
  Arms: SGLT 2 inhibitor

SUMMARY:
The aim of study is impact of additional treatment with new antidiabetic drugs (semaglutide or empagliflozine) compared to control group in T1DM patients - impact on endothelial function measured by FMD and FPF, arterial stiffness - measured by PWV, inflammatory biomarkers, markers of oxidative stress and endothelial progenitor cells (CD 34+/VDRL2, CD 133+/VDRL2) and correlation with glucovariability or time in range, measured with CGM system.

ELIGIBILITY:
Inclusion Criteria:

* T1DM
* HbA1C<=9%
* prone to CGM system
* 20 - 70 years

Exclusion Criteria:

* HbA1C >9%,
* BMI<22,
* pregnancy or lactation,
* known hypersensitivity to study drug,
* malignant disease ( excluded >5 years disease free, bazocellular or planocellular ca of skin),
* liver cirrhosis child C,
* eGFR<60 ml/min,
* chronic inflammatory disease,
* proliferative diabetic rethinopathy,
* MEN or medullary thyroid cancer in familly,
* concomitant drugs with influence on glycemia and antiinflammatory influence (corticosteroids, immunosupresive therapy),
* Major cardiovascular event last 2 months ( stroke, MI)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
evaluation of endothelial function by flow mediated dilation (FMD) of brachial artery | 12 weeks
  measurement of dilation of brachial artery (in %) before and after postishemic hyperemia comparing two therapeutic groups and control group before and after intervention
evaluation of endothelial function by strain gauge plethysmography as change in forearm blood flow | 12 weeks
  changes in tissue perfusion (ml/100 ml of tissue/min) measured with strange gauge plethysmography as formarm blood flow before and after postishemic reactive hyperemija comparing two therapeutic groups and control group before and after intervention
evaluation of arterial stiffness with peak wave velocity ( PWV) | 12 weeks
  measurements of the velocity (m/s) at which arterial blood pressure pulses propagate - comparing two therapeutic groups and control group before and after intervention

SECONDARY OUTCOMES:
evaluation of change in inflammatory biomarkers | 12 weeks
  change of hs CRF, Il6 after treatment comparing two therapeutic groups and control
evaluation of change in biomarkers of endothelial dysfunction | 12 weeks
  change in s-VCAM, s-ICAM values before and after intervention - comparing two therapeutic groups and control
evaluation of endothelial progenitor cells EPC count | 12 weeks
  change in count of endothelial progenitor cells CD 34*, 133+ as endothelial function markers before and after intervention - comparing two therapeutic groups and control

OTHER OUTCOMES:
body impedance measurements | 12 weeks
  changes in measurements of body composition fat , muscle and water before and after intervention - comparing two therapeutic groups and control
changes of glycemia endpoints glucovariability/time in range | 2 weeks
  variability of excursions of glucose - coeficient of variability / time in range defined as blood glucose beetwen 3,9 and 10 mmol/l before and after drug intervention assesed with CGM system

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, prof PhD, Study Chair — General and teaching hospital Celje and UKC Ljubljana/Maribor
Locations (1):
- General Hospital Celje, Celje, Slovenia

IPD SHARING:
Plan to Share IPD: No